CLINICAL TRIAL: NCT05840094
Title: A Prospective Study of the Predictive and Prognostic Value of Multimodalitic Imaging in the N-stage of Lung Cancer
Brief Title: Multimodalitic Imaging in the N-stage of Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCN001
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-03

CONDITIONS: Neoplasm of Lung
Keywords: 18F-FDG PET/CT; Neoplasm of Lung; EBUS-TBNA; MR STIR; NSCLC N-stage
MeSH Terms: conditions — Lung Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PET/CT+MR+EBUS (Experimental): Subjects will receive 18F-FDG PET/CT and MR STIR sequence combined with EBUS-TBNA, to diagnose the N-stage of NSCLC
  Interventions: Drug: 18F-FDG; Device: MR STIR; Procedure: EBUS-TBNA
- PET/CT+EBUS (Experimental): Subjects will receive 18F-FDG PET/CT and EBUS-TBNA, to diagnose the N-stage of NSCLC
  Interventions: Drug: 18F-FDG; Procedure: EBUS-TBNA
- MR+EBUS (Experimental): Subjects will receive 18F-FDG PET/CT and EBUS-TBNA, to diagnose the N-stage of NSCLC
  Interventions: Device: MR STIR; Procedure: EBUS-TBNA

INTERVENTIONS:
Drug: 18F-FDG — 18F-FDG is injected intravenously with a dose of 0.1mCi/kg.
  Arms: PET/CT+EBUS; PET/CT+MR+EBUS
Device: MR STIR — The overall scanning time of MR is about 13min.
  Arms: MR+EBUS; PET/CT+MR+EBUS
Procedure: EBUS-TBNA — Puncture about 20 times, 3 stitches in each group of enlarged lymph nodes, 1 stitch in the anterior, middle and posterior parts respectively

SUMMARY:
This study aims to evaluate the diagnostic efficacy and differences between 18F-FDG PET/CT and MR STIR sequences combined with EBUS-TBNA, 18F-FDG PET/CT combined with EBUS-TBNA, and MR STIR sequences combined with EBUS-TBNA - three types of multimodal imaging for assessing NSCLC N-stage, in order to select the best assessment protocol to guide treatment decisions and prognostic assessments.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy pathologically confirmed NSCLC, or clinically highly suspicious NSCLC (assessed as highly suspicious by the MDT team of this study);
* N1, N2, or N3 confined to the mediastinum and hilum, as assessed by imaging;
* Proposed systematic lymph node dissection without any treatment;
* Appropriate laboratory tests (serum tumor markers);
* All examination intervals ≤ 4 weeks;
* KPS score ≥ 50 (ECOG/WHO equivalent);
* Aged > 18 years; 8. Patients can fully understand and voluntarily participate in this trial and sign the informed consent; the examination can be completed independently.

Exclusion Criteria:

* Contraindication to EBUS-TBNA operation;
* Presence or history of other malignancies within 10 years;
* Inability to understand the examination procedure or to cooperate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The diagnostic efficacy of18F-FDG PET/CT and MR STIR sequences combined with EBUS-TBNA in the lymph node staging of NSCLC | 1 year
  Sensitivity, specificity, positive predictive value, negative predictive value, and accuracy of three multimodal methods for diagnosing mediastinal lymph node staging in NSCLC based on patients.

SECONDARY OUTCOMES:
The diagnostic efficacy of18F-FDG PET/CT combined with EBUS-TBNA in the lymph node staging of NSCLC | 1 year
  Sensitivity, specificity, positive predictive value, negative predictive value, and accuracy of two multimodal methods for diagnosing mediastinal lymph node staging in NSCLC based on patients.
The diagnostic efficacy of18F-FDG PET/CT combined with MR STIR in the lymph node staging of NSCLC | 1 year
  Sensitivity, specificity, positive predictive value, negative predictive value, and accuracy of two multimodal methods for diagnosing mediastinal lymph node staging in NSCLC based on patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided